CLINICAL TRIAL: NCT04203147
Title: HOME DM-BAT: Home-based Diabetes-Modified Behavioral Activation Treatment for Low Income Seniors With T2DM
Brief Title: Home-based Diabetes-Modified Behavioral Activation Treatment for Low Income Seniors With T2DM
Acronym: HOME DM-BAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R01DK118038-01A1 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-12-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home DM-BAT Intervention (Experimental): A trained nurse educator will deliver the manualized Home DM-BAT intervention. Subjects will receive 8-weekly sessions of behavioral activation and monthly booster sessions from months 3-12 via telephone.
  Interventions: Behavioral: Home DM-BAT
- Control Group (GHE+ST) (Active Comparator): Patients randomized to the control group will receive in-home 8-weekly sessions of combined general health education (GHE) and supportive therapy (ST) and monthly booster sessions from months 3-12 via telephone.
  Interventions: Behavioral: Supportive Therapy (Control)

INTERVENTIONS:
Behavioral: Supportive Therapy (Control) — Description: 8-weekly sessions of in-home, supportive therapy and monthly booster sessions from months 3-12 via telephone.
  Arms: Control Group (GHE+ST)
Behavioral: Home DM-BAT — Description: 8-weekly sessions of in-home, culturally-modified, manualized diabetes-modified, behavioral activation treatment (Home DM-BAT) and monthly booster sessions from months 3-12 via telephone.
  Arms: Home DM-BAT Intervention

SUMMARY:
The objective of this protocol is to evaluate the efficacy and cost-effectiveness of 8 sessions of in-home, telephone-delivered, culturally-modified, manualized diabetes-modified, behavioral activation treatment (Home DM-BAT) delivered by trained diabetes nurse educators among low income, ethnic minority seniors with poorly controlled T2DM.

The aims of this randomized controlled efficacy trial are:

Aim 1: To test the efficacy of Home DM-BAT on clinical outcomes (hemoglobin A1c, blood pressure, and LDL-Cholesterol).

Hypothesis 1: Low income, minority seniors with poorly controlled T2DM randomized to Home DM-BAT will have significantly greater improvements in clinical outcomes (hemoglobin A1c, blood pressure, and LDL-Cholesterol) at 12 months of follow-up compared to the control group (in-home, telephone-delivered supportive therapy - ST).

Aim 2: To test the efficacy of Home DM-BAT on behavioral outcomes (home blood glucose monitoring, diet, exercise and medication adherence) and quality of life.

Hypothesis 2: Low income, minority seniors with poorly controlled T2DM randomized to Home DM-BAT will have significantly greater improvements in behavioral outcomes (home blood glucose monitoring, diet, exercise and medication adherence) and quality of life (physical and mental health components of SF-12) at 12 months of follow-up compared to the control group.

Aim 3: To determine the cost-effectiveness of Home DM-BAT intervention for diabetes.

Hypothesis 3: Home DM-BAT will be more cost-effective in improving hemoglobin A1c levels at 12 months of follow-up, compared to the control group, as measured by differences in program costs, resource utilization, and hemoglobin A1c levels.

DETAILED DESCRIPTION:
Study Overview. Two hundred participants will be randomized 1:1 to Home DM-BAT (n=100) or the control condition (n=100) to control for attention. The intervention includes 8 weekly intervention sessions and 10 monthly booster sessions. Study assessments will be performed by blinded research assistants at baseline, 3-, 6-, 9-, and 12-months of follow-up. Primary analyses will be conducted at 12 months post-randomization.

Description of the Home DM-BAT Intervention: A trained nurse educator will deliver the manualized Home DM-BAT intervention via telephone. Subjects will receive 8-weekly sessions of behavioral activation and monthly booster sessions from months 3-12. All intervention sessions will be delivered by telephone and will include a previously tested diabetes education/skills training intervention based on ADA guidelines, diabetes-tailored behavioral activation and will address social determinant of health issues.

Control Group (GHE+ST): Patients randomized to the control group will receive in-home, telephone-delivered 8-weekly sessions of combined general health education (GHE) and supportive therapy (ST) and monthly booster sessions from months 3-12 to match the intervention group for both content and attention. The control group will not receive diabetes education, address social determinants of health, or behavioral activation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=65 years of age;
2. Self-identified as Black/African American or Hispanic;
3. Clinical diagnosis of T2DM verified by an HbA1c >=8% at the screening assessment;
4. Able to communicate in English or Spanish; and
5. Resident of independent, subsidized, assisted senior housing facility or community dwelling elderly adults in the greater Milwaukee area and surrounding counties that have high African American/Hispanic populations.

Exclusion Criteria:

1. Mental confusion at screening assessment suggesting significant dementia;
2. Participation in other diabetes research;
3. Alcohol or drug abuse/dependency;
4. Active psychosis or acute mental disorder; and
5. Life expectancy <12 months at screening assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | Change in baseline HbA1c at 12 months post intervention follow-up
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for HbA1c.
Systolic and Diastolic Blood Pressure | Change in baseline blood pressure at 12 months post intervention follow-up
  Blood pressure readings will be obtained using automated BP monitors (OMRON IntelliSenseTM HEM-907XL). The device will be programmed to take 3 readings at 2-minute intervals, and give an average of the 3 BP readings.
LDL-Cholesterol | Change in baseline cholesterol at 12 months post intervention follow-up
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for LDL-Cholesterol.

SECONDARY OUTCOMES:
Quality of Life as measured by SF-12 | Change in baseline quality of life measure at 12 months post intervention follow-up
  The SF-12 (Ware 1996) is a valid and reliable instrument to measure functional status and reproduces 90% of the variance in PCS-36 and MCS-36 scores.
Self-Care Behaviors | Change in baseline self-care behaviors at 12 months post intervention follow-up
  Behavioral skills will be assessed with the Summary of Diabetes Self-Care Activities (SDSCA) scale (Toobert 2000), a brief, validated questionnaire of diabetes self-care. Medication Adherence will be measured with the 6-item validated self-report Brooks Medication Adherence Scale (BMAS) (Brooks 1994). Each of 6 items measures a specific medication-taking behavior.

OTHER OUTCOMES:
Quality Adjusted Life Years as measured by EQ-5D | Change in baseline quality of life measure at 12 months post intervention follow-up
  The EQ-5D is a validated measure to assess health status developed by the EuroQol group, an international team of researchers. This scale assesses health status across 5 dimensions using 26 items (Herdman 2011).
Resource Utilization and Cost | Change in baseline baseline resource utilization and cost at 12 months post intervention follow-up
  Previously validated questions on resource utilization will be administered. The questionnaires capture information on hospitalizations, physician/professional visits, and medications.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Egede LE, Davidson TM, Knapp RG, Walker RJ, Williams JS, Dismuke CE, Dawson AZ. HOME DM-BAT: home-based diabetes-modified behavioral activation treatment for low-income seniors with type 2 diabetes-study protocol for a randomized controlled trial. Trials. 2021 Nov 8;22(1):787. doi: 10.1186/s13063-021-05744-1. PMID 34749788